CLINICAL TRIAL: NCT06885645
Title: A Phase 1 Study of KH815 for Injection to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity in Patients With Advanced Solid Tumors
Brief Title: First-In-Human Study in Participants With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KH815-30101
Record Dates: First submitted 2025-03-06; First posted 2025-03-20 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KH815 for Injection (Experimental): Phase I: Dose Escalation Phase I part of the study:dose1-dose5 of KH815 for injection
  Interventions: Drug: KH815 for injection

INTERVENTIONS:
Drug: KH815 for injection — KH815 for injection is a dual-payload Antibody Drug Conjugate (ADC) targeting TROP2 antigens.

SUMMARY:
A Phase 1 Study of KH815 for Injection to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
The study will use BOIN design for dosing cohort management to determine the MTD and RDE/RP2D. The starting dose of KH815 is 0.5 mg/kg, followed by 1.0 to 4.0 mg/kg. The investigational product will be administered on Day 1 every 3 weeks via intravenous infusion, and the first cycle of KH815 treatment is for DLT evaluation. Enrolled patients will be sequentially assigned to the planned dose levels as required by the protocol and treated with KH815 IV Q3W to observe the occurrence of treatment related AEs and dose limiting toxicities. The dose-escalation decision will be determined per discussion between Safety Review Committee and Sponsor if deemed necessary. Moreover, the SRC is also responsible for deciding the MTD and the recommended dose level for dose-expansion study.

ELIGIBILITY:
inclusion criteria:

1. Signed, written IRB-approved Informed Consent.
2. Male or female.
3. Aged 18 ~ 75 years.
4. Life expectancy of at least 3 months.
5. Histologically or cytologically confirmed advanced or unresectable solid tumors for wihch failure or difficult to be treated with standard therapies, or not suitable for standard therapies.
6. Measurable disease by CT/MRI as defined in RECIST v1.1.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.

exclusion criteria：

1. Pregnant or lactating women.
2. Received cancer-directed therapy within the following timeframes:

   * Major surgery within 4 weeks or will be expected to require major surgical treatment during the study period.
   * Radical radiotherapy or chest palliative radiotherapy within 4 weeks, or palliative radiotherapy at any other sites except chest within 2 weeks.
   * Antibody-based anti-cancer therapies, macromolecular protein products or cytotherapies within 4 weeks.
   * Hormonal anti-tumor therapy within 2 weeks.
   * Chemotherapy (including non-antibody based immunotherapy therapy) within 2 weeks (6 weeks for nitrosoureas or mitomycin C) or 5 times half life of the chemotherapeutic agent (whichever is longer).
   * Any natural medicine with anti-tumor effect within 2 weeks.
   * Tyrosine kinase inhibitor (TKI) treatment within 1 week.
3. Received experimental drug therapy or participated in a clinical study of a medical device within 4 weeks prior to first infusion of KH815.
4. Known history of unstable angina, myocardial infarction (MI), or congestive heart failure (CHF) (NYHA Class II-IV) within 6 months or clinically significant arrhythmia (other than stable atrial fibrillation or paroxysmal superventricular tachycardia) requiring anti-arrhythmia therapy
5. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) and/or diabetes (HbA1c ≥ 9.0%).
6. Uncontrolled pleural effusion or pericardial effusion. Ascites requiring repeated drainage surgery (once a month or more frequently).
7. Patients with moderate to severe respiratory dyspnea due to severe primary lung disease or complications of advanced malignancy [rated as grade 3/4 by modified Medical Research Council (mMRC) scale] (see Appendix 3), or requiring continuous oxygen therapy, or acute exacerbations of chronic obstructive pulmonary disease (AECOPD), or history of interstitial lung disease (ILD)/pneumonia, or ILD/ pneumonia that could not be ruled out on imaging during screening, or any autoimmune disease/connective tissue disease (e.g. Rheumatoid arthritis, Sjogren's syndrome, sarcoidosis) with lungs involvement.
8. Grade ≥2 anorexia, nausea, vomiting, or diarrhea within 2 weeks prior to first infusion of KH815.
9. Active central nervous system (CNS) metastasis (defined as untreated and has symptoms such as consciousness disorder, or need steroid or anticonvulsant therapy to control symptoms) within 1 month prior to first infusion of KH815.
10. History of significant active bleeding, intestinal obstruction, or gastrointestinal perforation within 6 months prior to first infusion of KH815.
11. Newly diagnosed thromboembolic events requiring treatment within 6 months prior to first infusion of KH815 [patients with controlled and stable lower extremity deep venous thrombosis (DVT) or catheter related thrombosis (CRT) could be included].
12. Known history of other malignancies diagnosed within 5 years prior to first infusion of KH815 (patients with basal cell carcinoma, skin squamous cell carcinoma and carcinoma in situ, and with radical resection for more than 3 years could be enrolled).
13. Known history of severe dry eye, severe meibomian gland disease or blepharitis, incurable or delayed corneal healing resulted from the keratopathy or macular disease.
14. Known to be allergic to any component of KH815, or known history of grade ≥3 anaphylaxis to macromolecular protein products/antibody-based therapy, or known history of grade ≥3 drug-related AEs with the use of topoisomerase I inhibitors such as irinotecan.
15. Patients who require use of strong inhibitors or inducers of CYP3A4 at least 14 days prior to the first infusion of KH815 and throughout study. Use of strong inhibitors or inducers of CYP3A4 is not allowed in this study.
16. Human immunodeficiency virus (HIV) antibody positive. Has an active or uncontrolled hepatitis B (HBV) and/or hepatitis C (HCV) infection. Patients with untreated or ongoing tuberculosis, but those who have undergone standard anti-tuberculosis treatment and have been confirmed as cured by the investigator could be included.
17. Known history of allogeneic cell or solid organ transplantation.
18. Active infection requiring systemic treatment within 2 weeks prior to the first infusion of KH815.
19. Live or live attenuated vaccine within 28 days prior to KH815 administration and live or live attenuated vaccine planned over the course of the study.
20. Known history of psychotropic substance abuse, alcohol abuse, or drug abuse.
21. Psychological, social, familial, or geographical factors that would prevent regular follow-up. Adults under guardianship, curatorship, safeguard of justice, or family empowerment measure are not eligible.
22. Otherwise considered inappropriate for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Postdose of last participant up to 12 months
  To determine the maximum tolerated dose (MTD)
Dose Limiting Toxicities (DLTs) | Baseline up to 21 days after the first dose
  To determine the Dose Limiting Toxicities (DLTs).
Recommended Doses for Expansion (RDEs) | Postdose of last participant up to 12 months
  To determine the recommended doses for expansion (RDEs).

SECONDARY OUTCOMES:
Cmax | Post last dose up to Day 60
  To characterize the Cmax of KH815-ADC, KH815 TAB, free Drug-E payload and free Drug-T payload.
Tmax | Post last dose up to Day 60
  To characterize the Tmax of KH815-ADC, KH815 TAB, free Drug-E payload and free Drug-T payload.
AUC0-t | Post last dose up to Day 60
  To characterize the AUC0-t of KH815-ADC, KH815 TAB, free Drug-E payload and free Drug-T payload.
AUCtau | Post last dose up to Day 60
  To characterize the AUCtau of KH815-ADC, KH815 TAB, free Drug-E payload and free Drug-T payload.
t1/2 | Post last dose up to Day 60
  To characterize the t1/2 of KH815-ADC, KH815 TAB, free Drug-E payload and free Drug-T payload.
Objective Response Rate (ORR) | Postdose of last participant up to 12 months
  To evaluate the objective response rate (ORR) of KH815 for injection when administered intravenously (IV) as monotherapy at the RDEs to patients with advanced solid tumors.
Phase I: ADA prevalence and incidence | Post last dose up to Day 60
  To assess the prevalence and incidence of anti-drug antibody (ADA) of KH815

IPD SHARING:
Plan to Share IPD: Yes